CLINICAL TRIAL: NCT02828046
Title: A Phase 1, Single Center, Randomized, Double-Blind, Placebo-Controlled, Single (Part 1) and Multiple (Part 2) Ascending Dose Study to Evaluate the Safety, Tolerability, PK and PD of M281 Administered to Healthy Volunteers
Brief Title: An Ascending Dose Study to Evaluate M281 Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MOM-M281-001
Record Dates: First submitted 2016-06-14; First posted 2016-07-11 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- M281 (Experimental): M281
  Interventions: Biological: M281

INTERVENTIONS:
Biological: M281
  Arms: M281
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, and PK/PD of M281 after single and multiple doses in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between 18 and 55 years, inclusive.
2. Good health
3. Body weight between 50 and 110 kg inclusive

Exclusion Criteria:

1. History of any drug allergy, hypersensitivity, or intolerance to any drug product that in the opinion of the Investigator would place the subject at particular risk and compromise the safety of the subject in the study.
2. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, psychiatric disease, or any other condition, that in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.
3. History or current diagnosis of substance dependence (except nicotine and caffeine) or alcohol abuse over the past 2 years, according to the criteria of DSM-IV-TR.
4. Smokes or has smoked more than 5 cigarettes per day in the last 90 days and is unable to stop smoking during in-patient observation period in clinic.
5. Unwillingness to abstain from alcohol for at least 24 hours prior to dosing with study medication until the time of discharge from the study unit and at least 24 hours prior to each ambulatory visit.
6. Plans to participate in another clinical trial while enrolled in this study and/or received an investigational drug and/or device within 60 days prior to admission.
7. Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days prior to admission.
8. History of splenectomy, asthma (with the exception of childhood asthma that has resolved), COPD, recurrent or current GI or respiratory infections.
9. On fluid restriction.
10. Systemic steroids within 3 months prior to the start of study drug administration, or any prescription medication(s) within 14 days of dose administration or any non-prescribed systemic or topical medication (including any herbal product) within 7 days prior to dose administration.
11. Vaccination within 1 month before dosing, or plans to receive vaccination during the study.
12. Any illness within 5 days, or clinically significant airway infections within 30 days, prior to first study drug dosing.
13. Positive urine drug screen (UDS) at screening.
14. Positivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Counts and Percentages of adverse events by treatment group | Baseline until up-to 12 weeks post-dose

SECONDARY OUTCOMES:
Serum concentrations of M281 will be summarized using descriptive statistics (arithmetic means, SDs, coefficients of variation, sample size, minimum, maximum, and geometric means). | Baseline up-to 12 weeks post-dose
PD of M281 will summarize changes in serum markers of inflammation. | Up until 12 weeks post dose

CONTACTS AND LOCATIONS:
Overall Officials: John Hogan, MPM, Study Director — Momenta Director of Clinical Operations; Tjerk Bosji, MD, Principal Investigator — PRA Research Physician
Locations (1):
- PRA Health Sciences, Zuidlaren, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided